CLINICAL TRIAL: NCT06091488
Title: Evaluation Of Clinical Results And Imaging Of Anterior Cruciate Ligament Reconstruction With Orthopure Xt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACL-PURE
Record Dates: First submitted 2023-10-11; First posted 2023-10-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: ACL; ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients with anterior cruciate ligament injury, in which the patient's own autologous tendons cannot be used, will be treated with the ligamentous reconstruction device.
  Interventions: Other: Orthopure

INTERVENTIONS:
Other: Orthopure — Reconstruction of the anterior cruciate ligament of the knee in the patient.

SUMMARY:
The purpose of this study is to evaluate subjective and objective clinical outcomes and imaging data of subjects undergoing reconstruction or revision of LCA reconstruction using OrthoPure XT

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 65 at the time of ACL reconstruction surgery;
* Patients aged 35 to 65 at the time of primary ACL reconstruction surgery;
* Male and female sex;
* First injury of the ACL with impossibility of use of autograft (patellar tendinopathy, quadriceps tendinopathy, goose leg tendinopathy) or refusal to use allograft (Bank tendon);
* Recurrence of ACL injury with impossibility of use of autograft (prior use/tendinopathy of the patellar, previous use/tendinopathy of the quadriceps, previous use/tendinopathy of the goose leg) or refusal to use allograft (tendon of Bank);

Exclusion Criteria:

* Patients who do not consent to be included in the study
* Presence of haematological, rheumatic or haemorrhagic disease time of assessment
* ACL primary reconstruction in subjects under 35
* Allergies and/or reactions from hypersensitivity or religious objection to the use of porcine derivation
* Pregnant and/or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee | At baseline (day 0)
  The score goes from 0 to 100 where the maximum is 100 and expresses the absence of limitations and symptoms, and therefore an excellent result; the further you go from this score and the worse the result, which can therefore be divided into four groups: excellent (80-100)good (60-80), good (30-60), bad (0-30)
International Knee Documentation Committee | After 2 months
  The score goes from 0 to 100 where the maximum is 100 and expresses the absence of limitations and symptoms, and therefore an excellent result; the further you go from this score and the worse the result, which can therefore be divided into four groups: excellent (80-100)good (60-80), good (30-60), bad (0-30)
International Knee Documentation Committee | After 6 months
  The score goes from 0 to 100 where the maximum is 100 and expresses the absence of limitations and symptoms, and therefore an excellent result; the further you go from this score and the worse the result, which can therefore be divided into four groups: excellent (80-100)good (60-80), good (30-60), bad (0-30)
International Knee Documentation Committee | After 24 months
  The score goes from 0 to 100 where the maximum is 100 and expresses the absence of limitations and symptoms, and therefore an excellent result; the further you go from this score and the worse the result, which can therefore be divided into four groups: excellent (80-100)good (60-80), good (30-60), bad (0-30)
Lysholm Knee Score | At baseline (day 0)
  The final score is obtained from the sum of the various scores obtained in the different and ranges from 0 to 100.
  Scores are divided into subgroups: Excellent (95-100); Good (84-94); Decent (65-83); Poor (<64).
Lysholm Knee Score | After 2 months
  The final score is obtained from the sum of the various scores obtained in the different and ranges from 0 to 100.
  Scores are divided into subgroups: Excellent (95-100); Good (84-94); Decent (65-83); Poor (<64).
Lysholm Knee Score | After 6 months
  The final score is obtained from the sum of the various scores obtained in the different and ranges from 0 to 100.
  Scores are divided into subgroups: Excellent (95-100); Good (84-94); Decent (65-83); Poor (<64).
Lysholm Knee Score | After 24 months
  The final score is obtained from the sum of the various scores obtained in the different and ranges from 0 to 100.
  Scores are divided into subgroups: Excellent (95-100); Good (84-94); Decent (65-83); Poor (<64).
Visual Analogue Scale | At baseline (day 0)
  is a one-dimensional quantitative pain assessment scale at 10 points; the scale requires the patient to select the number that best describes the intensity of his pain, from 0 to 10, at that precise moment. 0 means no pain and 10 indicates the worst possible pain.
Visual Analogue Scale | After 2 months
  is a one-dimensional quantitative pain assessment scale at 10 points; the scale requires the patient to select the number that best describes the intensity of his pain, from 0 to 10, at that precise moment. 0 means no pain and 10 indicates the worst possible pain.
Visual Analogue Scale | After 6 months
  is a one-dimensional quantitative pain assessment scale at 10 points; the scale requires the patient to select the number that best describes the intensity of his pain, from 0 to 10, at that precise moment. 0 means no pain and 10 indicates the worst possible pain.
Visual Analogue Scale | After 24 months
  is a one-dimensional quantitative pain assessment scale at 10 points; the scale requires the patient to select the number that best describes the intensity of his pain, from 0 to 10, at that precise moment. 0 means no pain and 10 indicates the worst possible pain.
Tegner Score | At baseline (day 0)
  allows to estimate the level of motor activity of a subject with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports
Tegner Score | After 2 months
  allows to estimate the level of motor activity of a subject with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports
Tegner Score | After 6 months
  allows to estimate the level of motor activity of a subject with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports
Tegner Score | After 24 months
  allows to estimate the level of motor activity of a subject with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports
continuity of the graft | After 24 months
  assess the continuity of the graft with magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Collins JE, Katz JN, Donnell-Fink LA, Martin SD, Losina E. Cumulative incidence of ACL reconstruction after ACL injury in adults: role of age, sex, and race. Am J Sports Med. 2013 Mar;41(3):544-9. doi: 10.1177/0363546512472042. Epub 2013 Jan 9. PMID 23302260
- [Result] Kessler MA, Behrend H, Henz S, Stutz G, Rukavina A, Kuster MS. Function, osteoarthritis and activity after ACL-rupture: 11 years follow-up results of conservative versus reconstructive treatment. Knee Surg Sports Traumatol Arthrosc. 2008 May;16(5):442-8. doi: 10.1007/s00167-008-0498-x. PMID 18292988
- [Result] Costa GG, Grassi A, Perelli S, Agro G, Bozzi F, Lo Presti M, Zaffagnini S. Age over 50 years is not a contraindication for anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2019 Nov;27(11):3679-3691. doi: 10.1007/s00167-019-05450-1. Epub 2019 Apr 3. PMID 30944945